CLINICAL TRIAL: NCT03031795
Title: Oral Ketorolac for Pain Relief During IUD Insertion: A Randomized Controlled Trial
Brief Title: Oral Ketorolac for Pain Relief During IUD Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OhioHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OH1-13-00503
Record Dates: First submitted 2016-11-30; First posted 2017-01-26 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Contraception
Keywords: intrauterine device
MeSH Terms: interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental (Experimental): ketorolac, oral, 20 mg, 1 dose, 45 minutes prior to IUD placement
  Interventions: Drug: Ketorolac
- placebo (Placebo Comparator): look alike placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac — Oral Tablet
  Other Names: Toradol
  Arms: experimental
Drug: Placebo — Oral Tablet
  Arms: placebo

SUMMARY:
Ketorolac is a non-steroidal anti-inflammatory drug (NSAID), similar to ibuprofen but it is used to treat more severe pain. Ketorolac (Trade name: Toradol) is typically used after surgical procedures. When taken orally, it should not cause sedation. The purpose of this study is to determine if oral ketorolac is effective at reducing pain during IUD placement versus a placebo tablet.

DETAILED DESCRIPTION:
In the United States, 10% of women choose an intrauterine device (IUD) for contraception. With typical use, unintended pregnancy rates in the first year of IUD contraception are 0.8% (Copper T) and 0.2% (LNG). It is known that long-acting, reversible contraception methods reduce the long-term cost of unintended pregnancies. A common deterrent to intrauterine contraception is the fear of pain during placement. Methods of pain relief during IUD insertion must be fast-acting but have minimal sedation. There have been many attempts to find effective pain relief during IUD placement. Neither ibuprofen nor naproxen have been shown to be effective in reducing pain. Misoprostol has been used to increase cervical ripening; however, pain was not decreased, and side effects of nausea and vomiting were increased. Ketorolac is a nonsteroidal anti-inflammatory drug (NSAID) that works by reversibly inhibiting cyclooxygenase-1 and 2.Time to peak plasma concentration ketorolac in the oral form is 44 minutes. Studies have shown that one dose of ketorolac can be as potent as morphine. Ketorolac is also well established for pain control in the immediate post-operative period. A recent study showed that intramuscular ketorolac wais effective in reducing pain after IUD insertion, but 20% of the participants reported that after the procedure, the injection site was as painful as the IUD placement. The current study was designed to evaluate if there is reduced pain during IUD placement using oral ketorolac 40-60 minutes before the procedure compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant
* English speaking women
* 18 years of age or older desiring an IUD for contraception

Exclusion Criteria:

* enrollment in another study
* pre-medication with any type of analgesic medication
* contraindication to an IUD
* weight under 50 kg
* allergy to non-steroidal anti-inflammatory medications
* past medical history of liver disease, renal disease, peptic ulcer disease or recent gastrointestinal bleed,
* daily narcotic pain use
* positive cultures for gonorrhea or chlamydia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Crawford, MD, Principal Investigator — OhioHealth

IPD SHARING:
Plan to Share IPD: No
We will share our published manuscript upon request:
  Crawford M, Davy S, Book N, Elliott JO, Arora A. Oral ketorolac for pain relief during intrauterine device insertion: a double-blinded randomized controlled trial. Journal of Obstetrics and Gynaecology Canada 2017, Dec;39(12):1143-1149. doi: 10.1016/j.jogc.2017.05.014.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: look alike placebo
  Placebos
Period: Overall Study
Arm/Group | Experimental | Placebo
Started | 35 | 36
Completed | 35 | 35
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ketorolac: Experimental group
- Placebo: Control group
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Placebo | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 36 | 71
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (6.7) | 30.7 (8.9) | 31.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: White | 27 | 22 | 49
  Race/ethnicity: Black | 5 | 10 | 15
  Race/ethnicity: Hispanic | 0 | 1 | 1
  Race/ethnicity: Asian | 1 | 1 | 2
  Race/ethnicity: Other | 2 | 2 | 4
  Race/ethnicity: Unknown | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 36 | 71

OUTCOME MEASURES:

1. Primary Outcome: Pain Before, During and After IUD Placement
Description: Pain before, during and after IUD placement on a 0 (no pain) to 10 (worst possible) scale. Higher score mean a worse outcome.
Time Frame: Before, during and after IUD placement
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo group
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 35 | 36
units on a scale
  Pain expected during the procedure | 4.1 (2.2) | 4.5 (2.4)
  Pre-procedure pain rating | 0.4 (1.0) | 0.7 (1.5)
  Tenaculum placement | 2.7 (2.2) | 3.2 (2.4)
  Uterine sounding | 3.3 (2.9) | 4.2 (2.9)
  Deployment of the IUD | 4.2 (2.9) | 5.7 (2.9)
  Overall pain rating during the procedure | 3.6 (2.9) | 4.9 (2.7)
  Level of pain 10 minutes post procedure | 1.1 (1.5) | 2.5 (2.5)
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; A 2 point difference was used to power the study. This is consistent with previous definitions of a clinically meaningful reductions in pain and provides a visually meaningful change on the 0-10 numerical rating scale with anchors at every other point, for example moving from "very severe" (8) to "severe pain" (6) or from "moderate pain" (4) to "mild pain" (2); Test type: Superiority; p < 0.05, Wilcoxon rank sum test — The a priori threshold for statistical significance was set at < 0.05 for each row comparison with no adjustment for multiple comparisons

ADVERSE EVENTS:
Time Frame: 45 minutes prior and up to 10 minutes post IUD placement
Arm/Group | Experimental | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No